CLINICAL TRIAL: NCT02611037
Title: A Phase 2 Study of Transarterial Chemoperfusion Treatment With Cisplatin, Methotrexate and Gemcitabine in Patients With Unresectable Pleural Mesothelioma
Brief Title: Transarterial Chemoperfusion: Cisplatin, Methotrexate, Gemcitabine for Unresectable Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18094
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Results first posted 2023-02-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Malignant Pleural Mesothelioma; Mesothelioma
Keywords: MPM; Unresectable; Respiratory; Intrathoracic; Transarterial; Chemoperfusion
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Cisplatin; Methotrexate; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemoperfusion + Questionnaire (Experimental): Transarterial Chemoperfusion treatment with cisplatin (35 mg/m^2), methotrexate (100 mg/m^2) and gemcitabine (1000 mg/m^2).
  Patients undergo angiogram and transarterial chemoperfusion treatment in every 4 weeks (3-6 weeks interval allowed) when cisplatin, methotrexate and gemcitabine will be administered into the thoracic aorta and/or the internal mammary artery on the side of the disease.
  Quality of life will be assessed using the modified version of the Lung Cancer Symptom Scale for Mesothelioma questionnaire.
  Interventions: Drug: Cisplatin; Drug: Methotrexate; Drug: Gemcitabine; Other: Lung Cancer Symptom Scale for Mesothelioma Questionnaire

INTERVENTIONS:
Drug: Cisplatin — The recommended dose of cisplatin for transarterial chemoperfusion in this study is 35 mg/m^2 body surface area (BSA). During the lead in phase of the study, 3 patients will be treated with regular doses of cisplatin.
  Other Names: Platinol
Drug: Methotrexate — The recommended dose of methotrexate for transarterial chemoperfusion in this study is 100 mg/m^2 BSA. During the lead in phase of the study, 3 patients will be treated with 50% reduced dose of methotrexate (50 mg/m^2).
  Other Names: Trexall; Rheumatrex
Drug: Gemcitabine — The recommended dose of gemcitabine for transarterial chemoperfusion in this study is 1000 mg/m^2 BSA. During the lead in phase of the study, 3 patients will be treated with regular doses of gemcitabine.
  Other Names: Gemzar
Other: Lung Cancer Symptom Scale for Mesothelioma Questionnaire — Quality of life will be assessed using the modified version of the Lung Cancer Symptom Scale for Mesothelioma questionnaire.
  Other Names: Quality of Life Assessment

SUMMARY:
The purpose of this study is to determine whether the transarterial chemoperfusion treatment with cisplatin, methotrexate and gemcitabine is safe and effective in adults with malignant pleural mesothelioma (MPM).

DETAILED DESCRIPTION:
This is an open-label, single arm, phase 2 study with a lead in safety cohort to evaluate the safety and efficacy of transarterial chemoperfusion treatment with cisplatin (35 mg/m2^), methotrexate (100 mg/m^2) and gemcitabine (1000 mg/m^2) in patients with unresectable MPM. During the lead in phase of the study, 3 patients will be treated with 50% reduced dose of methotrexate (50 mg/m^2) and regular doses of cisplatin (35 mg/m^2 body surface area (BSA)) and gemcitabine (1000 mg/m^2 BSA).

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed malignant pleural mesothelioma (MPM).
* Have unresectable MPM or the patient refuses surgery for resectable MPM.
* Have failed to respond first line standard of care chemotherapy or the patient refuses first line chemotherapy.
* Have measurable disease, by computed tomography (CT) or magnetic resonance imaging (MRI) per modified Response Evaluation Criteria in Solid Tumors (RECIST) for mesothelioma. Radiographic tumor assessment must be performed within 28 days prior to the first treatment.
* The predominant burden of disease lies in an arterial distribution which is accessible for transarterial chemoperfusion treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >60%).
* All baseline laboratory requirements will be assessed and should be obtained within 14 days of first treatment. Screening laboratory values must be met..
* Women participate in the study must be surgically sterile, post-menopausal, or women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation and after for a certain amount of time (up to 5 weeks) after the last treatment.
* Women must have a negative serum or urine pregnancy test within 24 hours prior to the start of transarterial chemoperfusion treatment.
* Men must be surgically sterile or must agree to use adequate contraception prior to study entry and for the duration of study participation and after for a certain amount of time (up to 14 weeks) after the last treatment.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must have signed and dated an Institutional Review Board (IRB) approved written informed consent form in accordance with regulatory and institutional guidelines.
* Must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, imaging studies, and other requirements of the study.
* This study permits the re-enrollment of a participant who has discontinued the study for a reason other than treatment failure or adverse event(s) of the study treatment.

Exclusion Criteria:

* Patients who have had chemotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Recovery means resolution to at least Grade 1 toxicity if there was no baseline toxicity or less than or equal to the patient's baseline value.
* May not be receiving any other investigational agents.
* Known brain metastases or leptomeningeal metastases. Patients with other extrapleural metastases are included in this study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin, methotrexate, gemcitabine or other agents used during the study. History of allergic reaction to intravenous iodinated contrast media is not contraindication to the study. Patients with history of mild allergic reaction to iodinated contrast media will be premedicated with 40 mg of prednisone by mouth (p.o.) 12 and 2 hrs before the transarterial chemoperfusion treatment to prevent allergic reaction. Patients with history of moderate and severe allergic reaction to iodinated contrast media or patients with history of mild allergic reaction to iodinated contrast media despite adequate premedication will undergo angiogram using carbon dioxide or a gadolinium based contrast agent.
* Uncontrolled intercurrent illness including, but not limited to, presence of other malignancy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or breastfeeding.
* HIV-positive patients receiving combination anti-retroviral therapy.
* Potential participants who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bela Kis, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoperfusion -Lead In: Transarterial Chemoperfusion treatment with cisplatin (35 mg/m^2), methotrexate (100 mg/m^2) and gemcitabine (1000 mg/m^2).
  Patients undergo angiogram and transarterial chemoperfusion treatment in every 4 weeks (3-6 weeks interval allowed) when cisplatin, methotrexate and gemcitabine will be administered into the thoracic aorta and/or the internal mammary artery on the side of the disease.
  Cisplatin: The recommended dose of cisplatin for transarterial chemoperfusion in this study is 35 mg/m^2 body surface area (BSA). During the lead in phase of the study, 3 patients will be treated with regular doses of cisplatin.
  Methotrexate: The recommended dose of methotrexate for transarterial chemoperfusion in this study is 100 mg/m^2 BSA. During the lead in phase of the study, 3 patients will be treated with 50% reduced dose of methotrexate (50 mg/m^2).
  Gemcitabine: The recommended dose of gemcitabine for transarterial chemoperfusion in this study is 1000 mg/m^2 BSA. During the lead in phase of the study, 3 patients will be treated with regular doses of gemcitabine.
- Chemoperfusion - Open Label: Transarterial Chemoperfusion treatment with cisplatin (35 mg/m^2), methotrexate (100 mg/m^2) and gemcitabine (1000 mg/m^2).
  Patients undergo angiogram and transarterial chemoperfusion treatment in every 4 weeks (3-6 weeks interval allowed) when cisplatin, methotrexate and gemcitabine will be administered into the thoracic aorta and/or the internal mammary artery on the side of the disease.
  Cisplatin: The recommended dose of cisplatin for transarterial chemoperfusion in this study is 35 mg/m^2 body surface area (BSA).
  Methotrexate: The recommended dose of methotrexate for transarterial chemoperfusion in this study is 100 mg/m^2 BSA.
  Gemcitabine: The recommended dose of gemcitabine for transarterial chemoperfusion in this study is 1000 mg/m^2 BSA.
Period: Overall Study
Arm/Group | Chemoperfusion -Lead In | Chemoperfusion - Open Label
Started | 7 | 27
Completed | 5 | 27
Not Completed | 2 | 0
Not completed — Withdrawal prior to treatment | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Chemoperfusion + Questionnaire: Transarterial Chemoperfusion treatment with cisplatin (35 mg/m^2), methotrexate (100 mg/m^2) and gemcitabine (1000 mg/m^2).
  Patients undergo angiogram and transarterial chemoperfusion treatment in every 4 weeks (3-6 weeks interval allowed) when cisplatin, methotrexate and gemcitabine will be administered into the thoracic aorta and/or the internal mammary artery on the side of the disease.
  Quality of life will be assessed using the modified version of the Lung Cancer Symptom Scale for Mesothelioma questionnaire.
  Cisplatin: The recommended dose of cisplatin for transarterial chemoperfusion in this study is 35 mg/m^2 body surface area (BSA). During the lead in phase of the study, 3 patients will be treated with regular doses of cisplatin.
  Methotrexate: The recommended dose of methotrexate for transarterial chemoperfusion in this study is 100 mg/m^2 BSA. During the lead in phase of the study, 3 patients will be treated with 50% reduced dose of methotrexate (50 mg/m^2).
  Gemcitabine: The recommended dose of gemcitabine for transarterial chemoperfusion in this study is 1000 mg/m^2 BSA. During the lead in phase of the study, 3 patients will be treated with regular doses of gemcitabine.
  Lung Cancer Symptom Scale for Mesothelioma Questionnaire: Quality of life will be assessed using the modified version of the Lung Cancer Symptom Scale for Mesothelioma questionnaire.
Arm/Group | Chemoperfusion + Questionnaire
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: Disease control rate of transarterial chemoperfusion treatment with cisplatin, methotrexate and gemcitabine in patients with unresectable malignant pleural mesothelioma using modified Response Evaluation Criteria in Solid Tumors (RECIST) for mesothelioma. DCR provided as percentage of participants with partial response + percentage of participants with stable disease.
Time Frame: Up to 3 years
Population: All evaluable participants. Study patients cannot be analyzed separately. No dose limiting toxicities observed, therefore all participants received same dosing.
Measure: Number; unit: percentage of participants
Arm/Group | Chemoperfusion + Questionnaire
Number analyzed (Participants) | 32
percentage of participants | 75

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined as the time from the first day of transarterial chemoperfusion treatment to death.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemoperfusion + Questionnaire
Number analyzed (Participants) | 32
months | 8.9 [5.7 to 15]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival defined as the time from the first day of transarterial chemoperfusion treatment to disease progression based on imaging findings using modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria for mesothelioma. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemoperfusion + Questionnaire
Number analyzed (Participants) | 32
months | 4.7 [2.5 to 7.4]

4. Secondary Outcome: Occurrence of Treatment Related Toxicity
Description: Safety was assessed by monitoring adverse events and serious adverse events; the association with study treatment was assessed, and severity graded using Common Terminology Criteria for Adverse Events (CTCAE) v.4.03. Number of events that were Possible, Probable or Definitely related to study treatment.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: related adverse events
Arm/Group | Chemoperfusion + Questionnaire
Number analyzed (Participants) | 32
related adverse events | 32

5. Secondary Outcome: Quality of Life Questionnaire Scores
Description: Quality of life will be assessed using the modified version of the Lung Cancer Symptom Scale for Mesothelioma questionnaire. Mesothelioma Symptom Scale includes 7 categories to rate on a scale of 1 to 10 regarding severity of symptoms during the last 24 hours. A higher number indicates more severe symptoms.
Time Frame: Up to 3 years
Population: Quality of life questionnaires were not collected, therefore this measure cannot be analyzed.
Arm/Group | Chemoperfusion + Questionnaire
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first day of treatment until 30 days after last date of treatment, an average of 7.8 months.
Groups:
- Chemoperfusion - Lead In: Transarterial Chemoperfusion treatment with cisplatin (35 mg/m^2), methotrexate (100 mg/m^2) and gemcitabine (1000 mg/m^2).
  Patients undergo angiogram and transarterial chemoperfusion treatment in every 4 weeks (3-6 weeks interval allowed) when cisplatin, methotrexate and gemcitabine will be administered into the thoracic aorta and/or the internal mammary artery on the side of the disease.
  Cisplatin: The recommended dose of cisplatin for transarterial chemoperfusion in this study is 35 mg/m^2 body surface area (BSA). During the lead in phase of the study, 3 patients will be treated with regular doses of cisplatin.
  Methotrexate: The recommended dose of methotrexate for transarterial chemoperfusion in this study is 100 mg/m^2 BSA. During the lead in phase of the study, 3 patients will be treated with 50% reduced dose of methotrexate (50 mg/m^2).
  Gemcitabine: The recommended dose of gemcitabine for transarterial chemoperfusion in this study is 1000 mg/m^2 BSA. During the lead in phase of the study, 3 patients will be treated with regular doses of gemcitabine.
Arm/Group | Chemoperfusion - Lead In | Chemoperfusion - Open Label
All-Cause Mortality (participants affected / at risk) | 2/5 | 21/25
Serious Adverse Events (participants affected / at risk) | 2/5 | 7/25
Other Adverse Events (participants affected / at risk) | 5/5 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoperfusion - Lead In (N=5) | Chemoperfusion - Open Label (N=25)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Dyspena (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (3)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoperfusion - Lead In (N=5) | Chemoperfusion - Open Label (N=25)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (11) | 16 (46)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (8) | 12 (33)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (7) | 8 (10)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 4 (12)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 3 (8)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 3 (7) | 12 (34)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 4 (5)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 12 (26)
Vomiting (Gastrointestinal disorders) | 0 (0) | 8 (8)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (6) | 7 (13)
Creatinine increased (Investigations) | 0 (0) | 5 (12)
INR increased (Investigations) | 2 (2) | 2 (6)
Alanine aminotransferase increased (Investigations) | 1 (2) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (2) | 2 (3)
White blood cell decreased (Investigations) | 0 (0) | 2 (5)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (6)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 8 (12)
Pain (General disorders) | 0 (0) | 4 (4)
Fever (General disorders) | 0 (0) | 2 (2)
Flu-like symptoms (General disorders) | 0 (0) | 2 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (3) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (3)
Blurred vision (Eye disorders) | 0 (0) | 2 (3)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT02611037/Prot_SAP_000.pdf